CLINICAL TRIAL: NCT03621436
Title: Clinical Evaluation of the Transcatheter Renal Venous Decongestion (TRVD™) System for Renal Venous Decongestion in Patients With Acute Decompensated Heart Failure (ADHF)
Brief Title: Clinical Evaluation of the TRVD™ System in ADHF
Acronym: TRVD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to sponsor decision
Sponsor: Magenta Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRD00202, DRD00208, DRD00214
Record Dates: First submitted 2018-06-14; First posted 2018-08-08 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Acute Heart Failure; Congestive Heart Failure; Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRVD Therapy (Experimental)
  Interventions: Device: TRVD Therapy

INTERVENTIONS:
Device: TRVD Therapy — A catheter-mounted expandable flow pump is to be deployed in a transfemoral venous catheterization procedure. Once in place, renal venous pressure is reduced to a pre-selected physiologic target pressure and kept there for up to 24 hours. After termination of TRVD therapy, the device is removed.

SUMMARY:
A prospective, multi-national, open-label clinical study which is conducted to asses the safety, feasibility and performance of the TRVD™ System in hospital-admitted patients with Acute Decompensated Heart Failure (ADHF) and evidence of reduced left ventricular ejection fraction.

The study will include patients who present with significant venous congestion, as evidenced by clinical, laboratory and imaging signs of fluid retention.

Study participation, for each enrolled subject, will last approximately 3 months post index procedure.

Patients will be evaluated from enrollment until hospital discharge, then at 30, 60, and 90 days post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older
2. Patient admitted to the hospital with a primary diagnosis of ADHF who is chronically treated with at least one oral loop diuretic.
3. Patient presents at least two of the following clinical signs of manifest volume overload: 3.1 Jugular venous distension 3.2 Dyspnea, rales, or evidence of pulmonary congestion or oedema on admission chest radiography 3.3 Abdominal discomfort compatible with internal organ congestion and/or hepatomegaly 3.4 Peripheral oedema
4. Ultrasonic evidence of IVC plethora, defined as IVC diameter >2.0 cm.
5. BNP levels >300 pg/dL or NT-proBNP >1500 pg/dL .
6. Evidence of cardiac etiology as per cardiac ultrasonography.
7. LVEF =/<40%.
8. CVP (Invasively measured) >/=14 mmHg
9. Male or non-pregnant / non-lactating female (NOTE: Females of child bearing potential must have a negative pregnancy test).
10. Patient understands the nature of the procedure and provides written informed consent prior to any study specific assessments.

Exclusion Criteria:

1. INR >3, use of a NOAC in the past 48 hours or contraindication to systemic anticoagulation with Heparin.
2. Evidence of hemodynamic instability, evidence of shock with organ hypoperfusion, or need for inotropic support.
3. Overt pulmonary oedema, or Respiratory insufficiency/hypoxia (peripheral haemoglobin saturation <90% with supplemental oxygen), need for non-invasive positive pressure ventilation or intubation.
4. Severe renal dysfunction (eGFR before decompensation <45 ml/min/1.73 m2 BSA or <25 on admission).
5. Known renal artery stenosis.
6. Known intrinsic kidney disease (e.g., established diagnosis of diabetic nephropathy with macroproteinuria, chronic glomerulonephritis).
7. Severe anaemia (haemoglobin <9 mg/dL).
8. Thrombocytopenia with a platelets count <100,000.
9. Acute coronary syndrome within 4 weeks prior to admission.
10. Active myocarditis or hypertrophic obstructive cardiomyopathy.
11. Complex congenital heart disease.
12. Severe valvular stenosis.
13. Severe morbid obesity (BMI >35).
14. Fluid retention that is not primarily of cardiac origin (e.g., advanced liver disease, severe hypo-albuminaemia, etc.)
15. Temperature > 38°C (oral or equivalent), or sepsis, or active systemic infection requiring IV anti-microbial treatment.
16. Large ascites per ultrasound/CT.
17. Cognitive impairment.
18. Planned PCI, or more than minor surgery in the next 3 months.
19. Moribund patient, or patient with malignancy or other comorbidities limiting life expectancy to less than one year.
20. Patient has a known allergy to Nickel.
21. Contraindication to recommended study medications or intravascular contrast material that cannot be adequately controlled with pre-medication.
22. Concurrent enrollment in another device or drug trial that has not completed the primary endpoint or clinically interferes with the current study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Preliminary Safety (device- and procedure-related SAEs) | 30 days post index procedure
  Incidence of device- and procedure-related SAEs
Feasibility (technical success) | Hospital discharge (at least 96 hours following index procedure)
  Rate of technical success (defined as successful delivery and deployment, adequate function during device operation and successful retrieval) at hospital discharge.
Feasibility (procedural success) | Hospital discharge (at least 96 hours following index procedure)
  Rate of procedural success (defined as absence of device-related SAEs) at hospital discharge.

SECONDARY OUTCOMES:
Initial performance (effectiveness of renal venous pressure reduction) | Up to 24 hours
  Invasively assessed renal venous pressure reduction from baseline (in mmHg)

CONTACTS AND LOCATIONS:
Locations (3):
- OLV-Hospital Aalst, Belgium, Aalst, Belgium
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Zemun Clinical Hospital Center, Belgrade, Serbia